CLINICAL TRIAL: NCT03700619
Title: Assessment of Executive Functions in Preterm Children in 11 to 12 Year Old From the Behavioral Rating Inventory of Executive Function (BRIEF) Questionnaire
Brief Title: Executive Functions and Preterm Children in 11 to 12 Year Old
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC18_0201
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Preterm Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: BRIEF parental survey — estimate incidence of executive functions disorders in preterm children in 11 to 12 year old, born less than 34 weeks of gestation, with the BRIEF parental questionnaire. Effects are potentially important because this study could objectify an increase of risk of executive functions disorders f in preterm children in 11 to 12 year old, and identify associated risk factors. This work could eventually alert pediatrician to be careful at the executive functions and to propose adapted supportive cares.

SUMMARY:
Preterm children have a high risk for neurodevelopmental impairments. The impact on motor functions and neurosensory functions is demonstrated but the incidence of executive functions is not described for preterm infants.

DETAILED DESCRIPTION:
It is an epidemiologic, observational, prospective study. All patients, included in the LIFT cohort, in 11 to 12 year old during the period study, are contacted by mail. Patients with congenital anomalies or genetic syndromes are excluded. Children with parents who do not speak French are excluded. Antenatal and postnatal criteria known to be associated with disorders of executive functions are collected as gestational age, sex, multiple pregnancy, intrauterine growth retardation, antenatal or postnatal steroid use, breastfeeding, cerebral injuries and socio-economic status. After a couple of weeks, parents are contacted by a study manager, by phone call, to collect parental consent and answer some parental questions. After consent collect, BRIEF questionnaires are sending. If they wish, parents could give the BRIEF teacher questionnaire to the mean teacher. Teachers send by themselves their response. An informatic version is available with a personal link given especially by mail for each child. All data are anonymous. BRIEF questionnaire is composed of 86 items, exploring 2 main domains: behavior and metacognition. Twenty minutes are necessary to complete questionnaire. In case of no questionnaire return after one month, parents are contacted by phone. The investigators hypothesize a lost to follow-up at 0.25 and no response at 0.35. The response expected is 300 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* patient in 11 to 12 year old, included in LIFT cohort

Exclusion Criteria:

* Congenital abnormalities including nervous system malformations; genetic diseases; incomplete understanding of written and oral French by parents

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients which former preterm of gestational age less than 34 weeks
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of disorders of executive functions in 11 to 12 year old in former preterm of gestational age less than 34 weeks, from the Behavioral Rating Inventory of Executive Function questionnaire. | 11 to 12 years after preterm birth.
  The sum of the 86 items is calculated.

SECONDARY OUTCOMES:
Find neonatal factors associated with executive functions disorders in former prematures in 11 to 12 year old | 11 to 12 years after preterm birth
  estimate adequacy between BRIEF questionnaire performed/completed by parents and BRIEF questionnaire performed by teacher.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France